CLINICAL TRIAL: NCT02716493
Title: Feasibility of an Eight-week Telerehabilitation Program for Patients With Unresectable Thoracic Neoplasia Receiving Chemotherapy
Brief Title: Feasibility of a 8-week Telerehabilitation Program for Patients With Thoracic Neoplasia Receiving Chemotherapy
Acronym: TELErp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Principal Investigator, Didier Saey, Dr, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 20994
Record Dates: First submitted 2016-03-10; First posted 2016-03-23 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Lung Cancer
Keywords: Telerehabilitation
MeSH Terms: conditions — Lung Neoplasms

ARMS (1):
- Telerehabilitation group (Experimental): Patients with unresectable thoracic neoplasia receiving chemotherapy treatment
  Interventions: Behavioral: Telerehabilitation program

INTERVENTIONS:
Behavioral: Telerehabilitation program — The intervention was an 8-week home-based telerehabilitation program (three sessions of about 75 minutes per week) using the eChez-Soi telerehabilitation platform.
  Through a unique software interface, the eChez-Soi allows for the following three technological aspects: 1- continuous data acquisition and recording from commercial biometric sensors; 2- continuous transmission of the collected data via the Internet to the clinician's computer, allowing the clinician to visualize the biomechanical and physiological parameters in real time; and 3- a challenging gaming environment with interactive exercises performed on musical rhythms.
  In total, 15 supervised sessions and 9 unsupervised sessions were planned for a total of 24 exercise sessions

SUMMARY:
Exercise-based rehabilitation improves physical function, fatigue and quality of life in patients with thoracic neoplasia. Consequently, the need for rehabilitation across the continuum of care in oncology is growing rapidly. However, the implementation of this type of intervention is limited because of many barriers such as patients' symptoms and poor accessibility to programs. In this context, healthcare systems should develop and implement new approaches to dispense these services. Consequently, telerehabilitation is a promising strategy to improve access and adherence to rehabilitation.

OBJECTIVES To investigate the feasibility, adherence and satisfaction of a home-based telerehabilitation program (TELERP) with real-time physiological parameters acquisition in patients with unresectable thoracic neoplasia receiving chemotherapy and to explore its effects on patients' functional capacity.

METHODS Five patients receiving chemotherapy followed an 8-week TELERP using real-time monitoring combined with interactive exercises. The TELERP included supervised (15) and unsupervised (9) strengthening and cardiovascular exercise sessions at a rate of 3 sessions/week. The feasibility of the TELERP, adverse outcomes, technical issues, program adherence and satisfaction were analysed. Prior to and after the program, a six-minute walking test (6MWT), a timed up and go (TUG) and a timed stair test (TST) were done to assess functional capacity

ELIGIBILITY:
Inclusion Criteria:

* Patients had to have an ECOG functional status of 0 (Asymptomatic) or 1 (Symptomatic but completely ambulatory);
* Have a sufficient understanding of verbal and written French instructions
* Live in a geographic region served by a high speed Internet connection.

Exclusion Criteria:

* oxygen pulsed saturation (SpO2) <80% during the cardiopulmonary exercise test
* contraindications to exercise testing according to the American Thoracic Society and American College of Chest Physicians Exercise Testing Guidelines
* cerebral or bone metastasis
* a history of significant cardiovascular disease, hypertension, diabetes or musculoskeletal concerns that might limit their ability to perform active exercises
* severe psychiatric illness compromising adherence to the rehabilitation training routine.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-11; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events during the 8-week telerehabilitation program | Along the 8-week program
Adherence of the participants to the 8-week telerehabilitation program. | Along the 8-week program
  Adherence was defined as the number of sessions done over the prescribed sessions (supervised and unsupervised) and as percentage of time spent within the target heart rate range (intensities) throughout the cardiovascular exercise sessions
Participants satisfaction with the telerehabilitation platform with the Québec User Evaluation of Satisfaction with Assistive Technology questionnaire (QUEST 2.0) | At the end of the 8-week telerehabilitation program
  The satisfaction of the patients was evaluated using a questionnaire adapted from the Québec User Evaluation of Satisfaction with Assistive Technology questionnaire (QUEST 2.0) that calculates both satisfaction scores for technological aspects and services. It consists of 12 items rated on a scale from 1 to 5 (1: not satisfied at all to 5: very satisfied).
User satisfaction with health services received with the French version of the Health Care Satisfaction Questionnaire | At the end of the 8-week telerehabilitation program
  To assess more specifically the user satisfaction with health services received, we used the French version of the Health Care Satisfaction Questionnaire. This is a 26-item questionnaire answered on a four-point Likert scale, where ''1'' represents ''not at all satisfied'' and ''4'' represents ''highly satisfied". The total score is calculated in percentage and can be computed as the mean overall satisfaction divided in three domains: i) relationship with the professional, ii) delivery of services and iii) organization of services. Higher scores indicate a higher level of satisfaction.

SECONDARY OUTCOMES:
Cardiopulmonary maximal exercise test (CPET) | At baseline and following the 8-week program
Constant workrate cycle exercise test at 80% of the maximal capacity of the patient | At baseline and following the 8-week program
Isokinetic quadriceps muscle functions | At baseline and following the 8-week program
  Quadriceps muscle function (strength and endurance) was assessed during an isokinetic endurance test performed at a rate of 30 repetitions at 90°/sec of angular velocity (Biodex, system pro 4, Biodex Medical System, 20 Ramsay Road, Shirley, New York )
Lean body mass | At baseline and following the 8-week program
  Lean body mass (in Kg) were measured by bioelectrical impedance analysis (TBF-300WA Tanita, Arlington Heights, IL, USA)
Fat body mass | At baseline and following the 8-week program
  Fat body mass (in Kg) were measured by bioelectrical impedance analysis (TBF-300WA Tanita, Arlington Heights, IL, USA)
Weight | At baseline and following the 8-week program
  Weight (in Kg) of the patient
Height | At baseline and following the 8-week program
  Height (in meters) of the patient
Timed up and go test | At baseline and following the 8-week program
Timed stairs test | At baseline and following the 8-week program
Distance achieved during the 6 minutes walking test | At baseline and following the 8-week program
Cancer specific quality of life with the self-reported European Organization for Research and Treatment of Cancer Quality of Life Questionnaire questionnaire | At baseline and following the 8-week program
  The cancer related quality of life was assessed using the self-reported European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-30) including the lung cancer specific questionnaire QLQ-LC13
Anxiety and depression with the Hospital Anxiety and Depression Scale questionnaire | At baseline and following the 8-week program
  The French Canadian version of the Hospital Anxiety and Depression Scale (HADS) was used to identify patients suffering of anxiety disorders or depression
Nutritional status with the mini-nutritional assessment | At baseline and following the 8-week program

CONTACTS AND LOCATIONS:
Locations (1):
- CRIUCPQ, Québec, Quebec, Canada